CLINICAL TRIAL: NCT01791348
Title: The Test-retest Effect of the "d2 Test of Attention" - a Test for Concentration and Performance.
Brief Title: The Test-retest Effect of the "d2 Test of Attention".
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Ilda Amirian, MD, PhD student, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: d2test_1234
Record Dates: First submitted 2013-02-06; First posted 2013-02-15 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Cognition and Attention in Surgeons and Nurses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- d2 test of attention (Other)
  Interventions: Other: d2 test of attention

INTERVENTIONS:
Other: d2 test of attention

SUMMARY:
The "d2 test of attention" has been used in studies regarding sleep deprivation due to night shifts in hospital staff, in order to determine whether sleep deprivation has an impact on performance. However, by repeating the test there appears to be a test-retest effect, as the participants improve when performing the test more than once. The aim of this study is to determine, whether the "d2 test of attention" has a test-retest effect.

DETAILED DESCRIPTION:
20 surgeons and 20 surgical nurses will be included in this study. They will be asked, after thorough instruction, to perform the d2 test of attention after a designed schedule. The participants will on day 1 and 2 perform the test 3 times consecutively at intervals of 5 minutes. On day 3, 4 and 5 the test will be repeated only once. After the 5th day follows a 7-day-break. On day 13 the test will again be performed once.

ELIGIBILITY:
Inclusion Criteria:

- Nurses and surgeons at the department of Surgery, Herlev hospital. Age 22-55 years.

Exclusion Criteria:

* Known sleep disturbances and attentional deficits, previous use of the d2 test of attention, use of central stimulating drugs

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Test score for the d2 test of attention | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jacon Rosenberg, MD, professor, chief surgeon,, Study Chair — Herlev Hospital, department of surgery, Herlev, Denmark
Locations (1):
- Herlev Hospital, department of surgery, Herlev, Denmark

REFERENCES:
- [Background] Niu SF, Chu H, Chen CH, Chung MH, Chang YS, Liao YM, Chou KR. A comparison of the effects of fixed- and rotating-shift schedules on nursing staff attention levels: a randomized trial. Biol Res Nurs. 2013 Oct;15(4):443-50. doi: 10.1177/1099800412445907. Epub 2012 May 15. PMID 22593230
- [Background] Bates ME, Lemay EP Jr. The d2 Test of attention: construct validity and extensions in scoring techniques. J Int Neuropsychol Soc. 2004 May;10(3):392-400. doi: 10.1017/S135561770410307X. PMID 15147597
- [Background] Schlosser K, Maschuw K, Kupietz E, Weyers P, Schneider R, Rothmund M, Hassan I, Bartsch DK. Call-associated acute fatigue in surgical residents--subjective perception or objective fact? A cross-sectional observational study to examine the influence of fatigue on surgical performance. World J Surg. 2012 Oct;36(10):2276-87. doi: 10.1007/s00268-012-1699-5. PMID 22752051